CLINICAL TRIAL: NCT01233609
Title: A Phase II Multiple Site, Randomized, Placebo-Controlled Trial of Oral Valproic Acid for Autosomal Dominant Retinitis Pigmentosa
Brief Title: Trial of Oral Valproic Acid for Retinitis Pigmentosa
Acronym: VPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Foundation Fighting Blindness (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-13371
Record Dates: First submitted 2010-11-01; First posted 2010-11-03 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Retinitis Pigmentosa
Keywords: retinitis pigmentosa; valproic acid; visual field
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valproic Acid (Active Comparator): Subjects who receive valproic acid
  Interventions: Drug: Valproic Acid
- Placebo (Placebo Comparator): Subjects who receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valproic Acid — One to four 250mg softgels by mouth daily (dose determined by body weight)
  Other Names: Valproate
  Arms: Valproic Acid
Drug: Placebo — Dosage per subject weight- same schedule as the active comparator
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate the efficacy of Valproic Acid (VPA) to both slow the progression of visual function loss and/or to restore visual function in patients with Autosomal Dominant Retinitis Pigmentosa (RP) and to collect safety and tolerability information.

DETAILED DESCRIPTION:
Retinitis Pigmentosa (RP) is an incurable and untreatable group of heterogeneous retinal degenerative diseases that cause severe visual loss. There is currently no therapeutic that substantially slows the progression of this disease, and certainly none that can restore vision in RP patients. The Valproic Acid (VPA) study is designed as a six-site, interventional, prospective, randomized, placebo controlled, double-blinded study of 90 participants to evaluate the efficacy of oral Valproic Acid to both slow the progression of visual function loss and/or to restore visual function in patients with an Autosomal Dominant RP genetic mutation and to collect safety and tolerability information. Patients that participate in the study will be randomized to either placebo or VPA in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Understand/sign the IRB-approved study informed consent document.
2. Age greater than or equal to 18 years, no upper age limit
3. Males and non-child bearing females must weigh ≥40 Kg and ≤158.9 Kg; Females of child bearing potential must weigh ≥40 Kg and ≤74.9 Kg.
4. Diagnosis of Retinitis Pigmentosa (RP).
5. Visual acuity of greater than or equal to 35 letters in at least one eye as measured by the EVA-ETDRS (equivalent to 20/200 on a Snellen chart).
6. Genotyped as autosomal dominant form of RP.
7. Female subjects of childbearing potential and male subjects able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must commit to practice at least two acceptable methods of contraception to minimize the chance of pregnancy during the study and for the 13 week period after stopping the study drug.
8. Female subjects of childbearing potential must have a negative urine pregnancy test at study entry and throughout the duration of the study.
9. Willingness to comply with the protocol.

Exclusion Criteria:

1. Medical problems that make consistent follow-up over the treatment period unlikely (e.g. stroke, severe MI, end stage malignancy), or in general a poor medical risk because of other systemic diseases or active uncontrolled infections.
2. Other retinal diseases: Glaucoma, retinal inflammatory disease (CME is allowable), cataract worse than +2 NS, or herpes simplex virus of the eye.
3. Intact visual field of 5⁰ or less.
4. Subject unable to provide reliable perimetry measurements in both eyes for both static and kinetic visual field, as determined by the Reading Center.
5. Diabetes.
6. History of cancer (other than non-melanoma skin cancer) diagnosed, or requiring treatment within the past 2 years.
7. A hemoglobin concentration, a platelet count or an absolute neutrophil count below the lower limit of normal at study entry.
8. Suspected liver dysfunction determined by having liver function values elevated above the upper limit of normal.
9. History of pancreatitis by clinical features and/or laboratory abnormalities in the last 12 months.
10. Renal dysfunction based on serum creatinine,(MDRD) equation.
11. Urea cycle disorders.
12. History of neurological conditions including epilepsy, history of brain injury, encephalitis, or any organic brain syndrome.
13. History of schizophrenia, schizoaffective disorder, bipolar disorder, suicidality or organic mental disorders.
14. Currently receiving valproic acid or other anti-convulsants.
15. Sensitive to or have ever had an allergic reaction to valproic Acid.
16. Sensitive to or have ever had an allergic reaction to peanuts as peanut oil is an inactive ingredient in valproic acid capsules and the placebo.
17. Has taken one of the disallowed drugs at least 2 weeks prior to randomization.
18. Pregnant women.
19. Lactating mothers who are breast feeding their babies.
20. RP patients involved in other clinical trials within the last 3 months.
21. Require enrollment by consent of a legally authorized representative.
22. Persons who are unable to read are not allowed to consent for themselves or others to participate in this study.
23. The potential participant lives in the same household as a current participant in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Zilliox, PhD, Study Director — Foundation Fighting Blindness
Locations (6):
- United States (6):
  - University of Miami, Bascom Palmer Eye Institute, Miami, Florida
  - University of Michigan, Ann Arbor, Ann Arbor, Michigan
  - Oregon Health & Science University, Portland, Oregon
  - University of Tennessee, Hamilton Eye Institute, Memphis, Tennessee
  - Retina Foundation of the Southwest, Dallas, Texas
  - University of Utah School of Medicine, Moran Eye Center, Salt Lake City, Utah

REFERENCES:
- [Background] Berson EL, Rosner B, Weigel-DiFranco C, Dryja TP, Sandberg MA. Disease progression in patients with dominant retinitis pigmentosa and rhodopsin mutations. Invest Ophthalmol Vis Sci. 2002 Sep;43(9):3027-36. PMID 12202526
- [Background] Bryant AE 3rd, Dreifuss FE. Valproic acid hepatic fatalities. III. U.S. experience since 1986. Neurology. 1996 Feb;46(2):465-9. doi: 10.1212/wnl.46.2.465. PMID 8614514
- [Background] Berson EL, Sandberg MA, Rosner B, Birch DG, Hanson AH. Natural course of retinitis pigmentosa over a three-year interval. Am J Ophthalmol. 1985 Mar 15;99(3):240-51. doi: 10.1016/0002-9394(85)90351-4. PMID 3976802
- [Background] Chen PS, Wang CC, Bortner CD, Peng GS, Wu X, Pang H, Lu RB, Gean PW, Chuang DM, Hong JS. Valproic acid and other histone deacetylase inhibitors induce microglial apoptosis and attenuate lipopolysaccharide-induced dopaminergic neurotoxicity. Neuroscience. 2007 Oct 12;149(1):203-12. doi: 10.1016/j.neuroscience.2007.06.053. Epub 2007 Jul 28. PMID 17850978
- [Background] Delyfer MN, Leveillard T, Mohand-Said S, Hicks D, Picaud S, Sahel JA. Inherited retinal degenerations: therapeutic prospects. Biol Cell. 2004 May;96(4):261-9. doi: 10.1016/j.biolcel.2004.01.006. PMID 15145530
- [Background] Dragunow M, Greenwood JM, Cameron RE, Narayan PJ, O'Carroll SJ, Pearson AG, Gibbons HM. Valproic acid induces caspase 3-mediated apoptosis in microglial cells. Neuroscience. 2006 Jul 21;140(4):1149-56. doi: 10.1016/j.neuroscience.2006.02.065. PMID 16600518
- [Background] Gaby AR. Nutritional therapies for ocular disorders: Part Three. Altern Med Rev. 2008 Sep;13(3):191-204. PMID 18950246
- [Background] Gottlicher M, Minucci S, Zhu P, Kramer OH, Schimpf A, Giavara S, Sleeman JP, Lo Coco F, Nervi C, Pelicci PG, Heinzel T. Valproic acid defines a novel class of HDAC inhibitors inducing differentiation of transformed cells. EMBO J. 2001 Dec 17;20(24):6969-78. doi: 10.1093/emboj/20.24.6969. PMID 11742974
- [Background] Hartong DT, Berson EL, Dryja TP. Retinitis pigmentosa. Lancet. 2006 Nov 18;368(9549):1795-809. doi: 10.1016/S0140-6736(06)69740-7. PMID 17113430
- [Background] Henry TR. The history of valproate in clinical neuroscience. Psychopharmacol Bull. 2003;37 Suppl 2:5-16. PMID 14624229
- [Background] Hoffman DR, Locke KG, Wheaton DH, Fish GE, Spencer R, Birch DG. A randomized, placebo-controlled clinical trial of docosahexaenoic acid supplementation for X-linked retinitis pigmentosa. Am J Ophthalmol. 2004 Apr;137(4):704-18. doi: 10.1016/j.ajo.2003.10.045. PMID 15059710
- [Background] Jacobson SG, Cideciyan AV, Huang Y, Hanna DB, Freund CL, Affatigato LM, Carr RE, Zack DJ, Stone EM, McInnes RR. Retinal degenerations with truncation mutations in the cone-rod homeobox (CRX) gene. Invest Ophthalmol Vis Sci. 1998 Nov;39(12):2417-26. PMID 9804150
- [Background] Kim HJ, Rowe M, Ren M, Hong JS, Chen PS, Chuang DM. Histone deacetylase inhibitors exhibit anti-inflammatory and neuroprotective effects in a rat permanent ischemic model of stroke: multiple mechanisms of action. J Pharmacol Exp Ther. 2007 Jun;321(3):892-901. doi: 10.1124/jpet.107.120188. Epub 2007 Mar 19. PMID 17371805
- [Background] Mangione CM, Lee PP, Gutierrez PR, Spritzer K, Berry S, Hays RD; National Eye Institute Visual Function Questionnaire Field Test Investigators. Development of the 25-item National Eye Institute Visual Function Questionnaire. Arch Ophthalmol. 2001 Jul;119(7):1050-8. doi: 10.1001/archopht.119.7.1050. PMID 11448327
- [Background] Noorwez SM, Ostrov DA, McDowell JH, Krebs MP, Kaushal S. A high-throughput screening method for small-molecule pharmacologic chaperones of misfolded rhodopsin. Invest Ophthalmol Vis Sci. 2008 Jul;49(7):3224-30. doi: 10.1167/iovs.07-1539. Epub 2008 Mar 31. PMID 18378578
- [Background] Nowomiejska K, Vonthein R, Paetzold J, Zagorski Z, Kardon R, Schiefer U. Comparison between semiautomated kinetic perimetry and conventional Goldmann manual kinetic perimetry in advanced visual field loss. Ophthalmology. 2005 Aug;112(8):1343-54. doi: 10.1016/j.ophtha.2004.12.047. PMID 15996734
- [Background] Nowomiejska K, Vonthein R, Paetzold J, Zagorski Z, Kardon R, Schiefer U. Reaction time during semi-automated kinetic perimetry (SKP) in patients with advanced visual field loss. Acta Ophthalmol. 2010 Feb;88(1):65-9. doi: 10.1111/j.1755-3768.2008.01407.x. Epub 2009 Dec 16. PMID 19094165
- [Background] Peterson GM, Naunton M. Valproate: a simple chemical with so much to offer. J Clin Pharm Ther. 2005 Oct;30(5):417-21. doi: 10.1111/j.1365-2710.2005.00671.x. No abstract available. PMID 16164485
- [Background] Wong R, Khan J, Adewoyin T, Sivaprasad S, Arden GB, Chong V. The ChromaTest, a digital color contrast sensitivity analyzer, for diabetic maculopathy: a pilot study. BMC Ophthalmol. 2008 Aug 17;8:15. doi: 10.1186/1471-2415-8-15. PMID 18706104
- [Derived] Birch DG, Bernstein PS, Iannacone A, Pennesi ME, Lam BL, Heckenlively J, Csaky K, Hartnett ME, Winthrop KL, Jayasundera T, Hughbanks-Wheaton DK, Warner J, Yang P, Fish GE, Teske MP, Sklaver NL, Erker L, Chegarnov E, Smith T, Wahle A, VanVeldhuisen PC, McCormack J, Lindblad R, Bramer S, Rose S, Zilliox P, Francis PJ, Weleber RG. Effect of Oral Valproic Acid vs Placebo for Vision Loss in Patients With Autosomal Dominant Retinitis Pigmentosa: A Randomized Phase 2 Multicenter Placebo-Controlled Clinical Trial. JAMA Ophthalmol. 2018 Aug 1;136(8):849-856. doi: 10.1001/jamaophthalmol.2018.1171. PMID 29879277
- See also: Click here for more information about this study: Clinical Trial page of the Foundation Fighting Blindness Website. — http://www.blindness.org/index.php?option=com_content&view=section&id=7&itemid=101

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valproic Acid | Placebo
Started | 46 | 44
Completed | 37 | 42
Not Completed | 9 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Valproic Acid | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (10.9) | 49.3 (12.3) | 50.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 44
  Male | 24 | 22 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 38 | 41 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 43 | 44 | 87
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Genetic Mutations [Count of Participants; unit: Participants] — Summary of participants' gene mutation or combination of mutations identified and thought to be responsible for autosomal dominant retinitis pigmentosa
  Participants
    RHO | 22 | 19 | 41
    PRPF31 | 5 | 9 | 14
    RP1 | 4 | 9 | 13
    PRPF8 | 3 | 1 | 4
    PRPH2 | 2 | 2 | 4
    NR2E3 | 0 | 2 | 2
    RHO and PRPH2 | 2 | 0 | 2
    SNRNP200/ASCC3L1 | 2 | 0 | 2
    TOPORS | 0 | 2 | 2
    IMPDH1 | 1 | 0 | 1
    KLHL7 | 1 | 0 | 1
    NR2E3 and TOPORS | 0 | 1 | 1
    RHO and ROM1 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Field Area From Baseline to 52 Weeks--III4e Isopter
Description: Mean change in visual field area from baseline to 52 weeks. Visual field area is measured with semi-automated kinetic perimetry (SKP) using the Octopus 900 (Haag-Streit) with the III4e target size for each eye and done at least twice to ensure reliable sessions; the visual field area measurements are averaged over the two sessions. Analysis performed with linear mixed model
Time Frame: baseline to week 52
Population: The analysis followed the intent-to-treat principle in that all randomized participants were included and analyzed according to their treatment assignment regardless of amount or type of treatment received. Only observed data were analyzed.
Measure: Mean (Standard Deviation); unit: Visual field area (degrees squared)
Units Other Than Participants: eyes
Groups:
- Placebo--Right Eye: Right eye of Placebo-treated patients
- Placebo--Left Eye: Left eye of Placebo-treated patients
- Valproic Acid--Right Eye: Right eye of Valproic acid-treated patients
- Valproic Acid--Left Eye: Left eye of Valproic acid-treated patients
Arm/Group | Placebo--Right Eye | Placebo--Left Eye | Valproic Acid--Right Eye | Valproic Acid--Left Eye
Number analyzed (Participants) | 42 | 42 | 38 | 38
Number analyzed (eyes) | 42 | 42 | 38 | 38
Visual field area (degrees squared) | -122.9 (543.60) | -112.0 (584.63) | -293.7 (736.56) | -237.1 (691.76)
Statistical Analysis 1: Comparison: Placebo--Right Eye vs Placebo--Left Eye vs Valproic Acid--Right Eye vs Valproic Acid--Left Eye; Test type: Superiority; p = 0.035, Mixed Models Analysis; degrees of freedom = 830; Mean Difference (Net) = -150.43, Standard Error of Mean 71.37 — Right eye and Left Eye within each of the 2 treatment groups (Placebo and Valproic Acid) were combined to estimate the difference

2. Secondary Outcome: Mean Change in Visual Field Area From Baseline to 52 Weeks--I4e Isopter
Description: Mean change in visual field area from baseline to 52 weeks. Visual field area is measured with semi-automated kinetic perimetry (SKP) using the Octopus 900 (Haag-Streit) with the I4e target size for each eye and done at least twice to ensure reliable sessions; the visual field area measurements are averaged over the two sessions. Analysis performed with linear mixed model
Time Frame: baseline to week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Visual field area (degrees squared)
Units Other Than Participants: eyes
Arm/Group | Placebo--Right Eye | Placebo--Left Eye | Valproic Acid--Right Eye | Valproic Acid--Left Eye
Number analyzed (Participants) | 42 | 42 | 38 | 38
Number analyzed (eyes) | 42 | 42 | 38 | 38
Visual field area (degrees squared) | 80.9 (406.2) | 115.7 (696.89) | 5.3 (759.46) | 19.5 (703.83)
Statistical Analysis 1: Comparison: Placebo--Right Eye; Test type: Superiority; p = 0.581, Mixed Models Analysis

3. Secondary Outcome: Static Perimetry by Treatment Arm--Full Field Hill of Vision
Description: Mean change from baseline at week 52 for Full field Hill of Vision (Static perimetry)
Time Frame: baseline to week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: db-steridians
Units Other Than Participants: eyes
Arm/Group | Placebo--Right Eye | Placebo--Left Eye | Valproic Acid--Right Eye | Valproic Acid--Left Eye
Number analyzed (Participants) | 41 | 41 | 39 | 39
Number analyzed (eyes) | 41 | 41 | 39 | 39
db-steridians | -0.3 (2.55) | -1.4 (3.27) | -0.2 (5.11) | -0.6 (4.68)
Statistical Analysis 1: Comparison: Placebo--Right Eye; Test type: Superiority; p = 0.409, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Static Perimetry Volume--30 Degree Hill of Vision
Description: Mean Change from baseline to week 52 for Static Perimetry Volume --30 Degree Hill of Vision. Full field static perimetry protocol was followed using the Octopus 900 (Haag-Streit) for a single session for each eye.
Time Frame: baseline to week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: db-steridans
Units Other Than Participants: eyes
Arm/Group | Placebo--Right Eye | Placebo--Left Eye | Valproic Acid--Right Eye | Valproic Acid--Left Eye
Number analyzed (Participants) | 41 | 41 | 39 | 39
Number analyzed (eyes) | 41 | 41 | 39 | 39
db-steridans | -0.3 (0.61) | -0.3 (0.73) | -0.2 (1.07) | -0.2 (0.96)
Statistical Analysis 1: Comparison: Placebo--Right Eye; Test type: Superiority; p = 0.229, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity
Description: Mean change in best corrected visual acuity as assessed by ETDRS (Early Treatment Diabetic Retinopathy Study) method from baseline to week 52
Time Frame: baseline to week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters read correctly
Groups:
- Valproic Acid -- Right Eye: Results from the Right Eye in Patients treated with Valproic Acid
- Valproic Acid--Left Eye: Results from the Left Eye in Patients treated with Valproic Acid
- Placebo --Right Eye: Results from the Right Eye in Patients treated with Placebo
- Placebo --Left Eye: Results from the Left Eye in Patients treated with Placebo
Arm/Group | Valproic Acid -- Right Eye | Valproic Acid--Left Eye | Placebo --Right Eye | Placebo --Left Eye
Number analyzed (Participants) | 40 | 40 | 42 | 42
letters read correctly | -1.4 (5.21) | 0.0 (3.41) | 0.2 (4.41) | 1.3 (5.05)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events are defined as those that occur between the first dose of study drug and the last dose of study drug plus 7 days.
Arm/Group | Placebo | Valproic Acid
All-Cause Mortality (participants affected / at risk) | 0/44 | 1/46
Serious Adverse Events (participants affected / at risk) | 2/44 | 3/46
Other Adverse Events (participants affected / at risk) | 41/44 | 45/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | Valproic Acid (N=46)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Road Traffic Accidents (Injury, poisoning and procedural complications) | 0 | 1 — Motorcycle crash
Immunodeficiency common variable (Immune system disorders) | 0 | 1 — Common Variable Immune Deficiency
Lens Dislocation (Eye disorders) | 1 | 0
Atrial Fibrilation (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | Valproic Acid (N=46)
Nasopharyngitis (Infections and infestations) | 9 | 3
Sinusitis (Infections and infestations) | 3 | 7
Influenza (Infections and infestations) | 7 | 1
Bronchitis (Infections and infestations) | 0 | 3
Nausea (Gastrointestinal disorders) | 3 | 8
Dyspepsia (Gastrointestinal disorders) | 0 | 8
Diarrhea (Gastrointestinal disorders) | 1 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 3
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 3
Vision Blurred (Eye disorders) | 5 | 3
Cystoid Macular Oedema (Eye disorders) | 1 | 3
Ammonia Increased (Investigations) | 1 | 7
Alanine Aminotransferase Increased (Investigations) | 2 | 3
Aspartate Aminotransferase Increased (Investigations) | 1 | 3
Weight Increased (Investigations) | 0 | 4
Hepatic Enzyme Increased (Investigations) | 0 | 3
Headache (Nervous system disorders) | 4 | 8
Dizziness (Nervous system disorders) | 3 | 2
Tremor (Nervous system disorders) | 0 | 3
Fatigue (General disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No